CLINICAL TRIAL: NCT03344094
Title: Mechanism of Action of Ocrelizumab in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB10681A
Record Dates: First submitted 2017-10-13; First posted 2017-11-17 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis; Immune System Diseases
MeSH Terms: conditions — Multiple Sclerosis; Immune System Diseases | interventions — ocrelizumab; Interferon-beta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — frozen cells and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- MS-ocrelizumab treated: ocrelizumab 600 mg IV over 5 hours, twice a year, with loading dose of 300 mg 2 weeks apart x 2 at start
  Interventions: Drug: ocrelizumab
- MS untreated: age- and sex-matched untreated MS controls
- Healthy control: age- and sex-matched untreated healthy controls
- MS interferon-treated: MS with ongoing interferon-beta therapy

INTERVENTIONS:
Drug: ocrelizumab — FDA-approved MS drugs
  Other Names: interferon-beta
  Groups: MS-ocrelizumab treated

SUMMARY:
Ocrelizumab is FDA approved for therapy of multiple sclerosis (MS). It depletes B cells and stops MS inflammation.

DETAILED DESCRIPTION:
The study will investigate immune cell subsets, and how the cells are modified by this therapy over a 1-year period in 25 subjects. Blood will be drawn at baseline, 2 weeks, 6 mo, and 12 mo.

Immune subsets will be analyzed by flow cytometry. Data are analyzed with ANOVA with repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are eligible for Ocrelizumab therapy based on FDA criteria

Exclusion Criteria:

* All patients who are ineligible for Ocrelizumab therapy based on FDA criteria.
* Prior treatment with Alemtuzumab or stem cell therapy, or immune abnormalities that would interfere with planned tests.
* Hepatitis B and HIV infections.
* Pregnant or lactating women.
* Hypersensitivity to trial medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MS and healthy controls from the U of Chicago Neurology Clinic population
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: anthony t reder, md, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: began 2-23-2018; filled 3-9-2018
Pre-assignment Details: not needed
Period: Overall Study
Arm/Group | MS-ocrelizumab Treated | MS Untreated | Healthy Control | MS Interferon-treated
Started | 15 | 5 (5) | 5 (5) | 5 (5)
Completed | 15 | 5 (5) | 5 (5) | 5 (5)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MS-ocrelizumab Treated | MS Untreated | Healthy Control | MS Interferon-treated | Total
Number analyzed (Participants) | 15 | 5 | 5 | 5 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 5 | 5 | 5 | 27
  >=65 years | 3 | 0 | 0 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (14.3) | 48.5 (14.8) | 55.1 (13.7) | 41.8 (2.5) | 48.4 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 1 | 3 | 18
  Male | 5 | 1 | 4 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 3 | 1 | 0 | 1 | 5
  White | 9 | 4 | 5 | 4 | 22
  More than one race | 2 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Chicago metropolitan area
  participants
    United States | 15 | 5 | 5 | 5 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Depletion of B Cells
Description: measured through lymphocyte surface marker stains, from patients, before and after ocrelizumab (Ocrevus) therapy Mononuclear cells (MNC) will be stained, for flow cytometry, with marker antibodies to B cells.
  The change in the percentage of each subset will be compared before and after treatment with paired t tests and ANOVA.
Time Frame: 1 year
Population: The MS-ocrelizumab treated group was analyzed for depletion of B cells, whereas MS-untreated, healthy controls and MS interferon-treated groups were not analyzed for depletion of B cells.
Measure: Count of Participants; unit: Participants
Groups:
- MS-ocrelizumab Treated: ocrelizumab 600 mg IV over 5 hours, twice a year, with loading dose of 300 mg 2 weeks apart x 2 at start
  ocrelizumab: FDA-approved MS drugs
  all enrolled
- MS Untreated: age- and sex-matched untreated MS controls
  all enrolled
- Healthy Control: age- and sex-matched untreated healthy controls
  all enrolled
- MS Interferon-treated: MS with ongoing interferon-beta therapy
  all enrolled
Arm/Group | MS-ocrelizumab Treated | MS Untreated | Healthy Control | MS Interferon-treated
Number analyzed (Participants) | 15 | 0 | 0 | 0
Participants | 15 | 0 | 0 | 0
Statistical Analysis 1: Comparison: MS-ocrelizumab Treated; Test type: Other — changes in subsets paired and unpaired t-tests, ANOVA; p = 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | MS-ocrelizumab Treated | MS Untreated | Healthy Control | MS Interferon-treated
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/15 | 0/5 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2010-01-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT03344094/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT03344094/ICF_001.pdf